CLINICAL TRIAL: NCT04829682
Title: Testing the Efficacy of ACT for Life: A Brief Inpatient Intervention to Maximize Recovery and Prevent Future Suicidal Behavior
Brief Title: Testing the Efficacy of ACT for Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3547-R; RX003547 (Other Grant/Funding Number: VA Rehabilitation Research and Development)
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Suicide
Keywords: Suicide; Inpatient; Veteran; Acceptance and Commitment Therapy; Present Centered Therapy
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to ACT for Life or Present Centered Therapy. Additionally all participants will continue to receive treatment as usual.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everyone except for the biostatistician will be blind to condition until randomization at the end of the pre-treatment assessment session. Outcome assessors will remain blind to condition for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT for Life (Experimental): ACT for Life + Treatment as Usual
  Interventions: Behavioral: ACT for Life
- Present Centered Therapy (Active Comparator): Present Centered Therapy + Treatment as Usual
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: ACT for Life — ACT for Life is a brief recovery oriented individual inpatient Acceptance and Commitment Therapy treatment protocol consisting of four modules typically administered in three to six inpatient sessions and one to four outpatient sessions in the 30 days following discharge from inpatient care. The immediate goals of ACT for Life are to increase the participant's psychological flexibility and readiness to cope effectively with future suicidal crises.
  Arms: ACT for Life
Behavioral: Present Centered Therapy — PCT is an evidence-based treatment for PTSD but its principles can be applied to psychotherapy for a wide range of difficulties. The standard PCT manual was originally adapted for suicide prevention by Craig Bryan and his colleagues. Our study team made additional minor revisions to prepare the manual for use as an active control condition in the current efficacy trial. PCT includes two initial sessions focused on discussion of current symptoms, psychoeducation, and the rationale for PCT. Current life problems become the focus of the remaining sessions. PCT is expected to consist of three to six, 60-90-minute inpatient sessions and one to four outpatient sessions in the 30 days following discharge. Discontinuation will occur when the participant attends an individual outpatient mental health appointment or 30 days after discharge, whichever occurs first. PCT participants will receive caring communications from their therapist for 12-months following inpatient discharge.
  Arms: Present Centered Therapy

SUMMARY:
Psychiatric hospitalization is a critical opportunity to provide treatment to reduce the risk of suicide and lay the groundwork for functional recovery. In fact, the period following psychiatric hospitalization presents the greatest risk of death by suicide for Veterans. Despite psychiatric hospitalization being a vital time for intervention, there are no suicide-specific evidence-based psychotherapies (EBPs) that can be feasibly delivered during a typical VHA inpatient stay. Importantly, suicide-specific inpatient interventions are primarily focused on reducing the reoccurrence of suicidal behavior and have limited or no focus on directly targeting other aspects of functional recovery. Preventing suicide during a crisis is only a short-term solution if we fail to assist patients in building a life they deem worth living.

The investigators' research over the past several years has been focused on addressing this gap and overcoming barriers to implementing psychosocial interventions in an inpatient setting. Acceptance and Commitment Therapy (ACT) is a psychosocial intervention well suited to both preventing suicide and enhancing functioning, but the investigators were not aware of any ACT-based treatment protocols designed to specifically target suicide risk. The investigators consulted with leading ACT clinicians and researchers to develop and manualize "ACT for Life", a brief, transdiagnostic, recovery-oriented, inpatient, intervention for Veterans hospitalized due to suicide risk. The individual intervention involves 3 to 6 inpatient sessions and 1 to 4 outpatient sessions focused on skills generalization and treatment engagement. The investigators conducted a randomized controlled pilot study evaluating the acceptability of ACT for Life and the feasibility of the planned design for the proposed randomized controlled efficacy trial. Results of this rigorous pilot study support the acceptability and feasibility of ACT for Life. Nearly all Veterans reported that they believed they benefitted from ACT for Life. Preliminary outcomes suggest that ACT for Life may improve functioning and reduce suicidal behavior following hospitalization due to suicide risk. However, a full-scale clinical trial will be necessary to definitively evaluate the efficacy of ACT for Life. To accomplish this goal, the investigators are proposing to conduct a randomized controlled trial of ACT for Life versus Present Centered Therapy in 278 Veterans hospitalized for suicide risk to examine outcomes of suicidal behavior and changes in functioning over a one-year period following psychiatric hospitalization. The specific aims of this study are to determine the efficacy of ACT for Life for preventing suicidal behavior and maximizing functional recovery, and to examine candidate ACT for Life treatment mechanisms. Participants will complete assessments prior to treatment, before discharge from the inpatient unit, and at one-, three-, six-, and twelve-months following discharge. The proposed randomized controlled trial of ACT for Life has the potential to fill the VHA's need for empirically-supported inpatient interventions that can be delivered during a typical inpatient stay, are recovery oriented, and prevent future suicidal behavior.

DETAILED DESCRIPTION:
Veterans are most likely to die by suicide in the week following discharge from acute psychiatric care. Brief, recovery-oriented, empirically-supported, inpatient interventions are needed given the unfortunate reality that Veterans at the greatest risk for suicide may not follow up with outpatient treatment. To effectively intervene on the many pathways to suicide, VHA will need to utilize brief inpatient psychosocial treatments that are suicide-specific and transdiagnostic. Acceptance and Commitment Therapy (ACT) is an evidence-based treatment approach ideally suited for utilization among Veterans at high risk for suicide because it simultaneously targets processes to reduce risk (e.g., distress tolerance) and to increase protective factors (e.g., engage patients in building a life they value). The ACT clinician does not focus on symptom reduction, but instead directly targets functional recovery by assisting patients in identifying and engaging in values-consistent behaviors even in the presence of aversive thoughts, emotions, or sensations. Furthermore, ACT is suitable for extremely brief interventions. ACT clinicians employ experiential exercises and metaphors that facilitate rapid new learning, and overcome many of the limitations of more verbally intensive, didactic approaches to therapy. Research studies in non-Veteran-specific populations indicate that as few as three ACT contact hours are associated with approximately 50% reductions in rehospitalization among patients with psychosis. The extant literature and qualities inherent to ACT strongly suggest that ACT could be effective for improving the functioning of Veterans at risk of suicide and in-turn preventing suicidal behavior; but these assumptions have yet to be empirically tested. To address this gap and overcome barriers to delivering targeted psychological interventions for suicide in a psychiatric inpatient setting, the investigators have developed and manualized a brief, transdiagnostic, recovery-oriented, suicide-specific, ACT intervention for Veterans hospitalized due to suicide risk, "ACT for Life". With the support of a Rehabilitation Research and Development (RR&D) Small Projects in Rehabilitation Research (SPiRE) grant the investigators conducted a randomized controlled acceptability and feasibility trial (N = 70), which demonstrated the acceptability of ACT for Life to Veterans hospitalized due to suicide risk. Data also support the feasibility of the proposed design for a full-scale randomized controlled trial evaluating the efficacy of ACT for Life for maximizing functioning after a suicidal crisis and preventing future suicidal behavior. Using a multisite, two arm, randomized controlled design (ACT for Life + Treatment as Usual [ACT] vs. Present Centered Therapy + Treatment as Usual [PCT]) with 278 participants, and assessments at pre-treatment, pre-inpatient-discharge, and one-, three-, six-, and 12-months post-inpatient-discharge, the investigators will:

Primary Aim: Determine the efficacy of ACT for Life for preventing suicidal behavior and maximizing functional recovery. Primary Hypothesis 1 is that ACT participants will be significantly less likely to engage in suicidal behavior (i.e., suicide or actual, aborted, or interrupted suicide attempts as assessed by the Columbia-Suicide Severity Rating Scale and medical record review) compared to PCT participants during the 12-months following psychiatric hospitalization. Primary Hypothesis 2 is that ACT participants will report significantly greater improvements in functioning on the Outcome Questionnaire 45.2 (OQ-45) compared to PCT participants at one-month post-discharge from psychiatric hospitalization.

Secondary Aims will examine onset and maintenance of treatment gains. Secondary Aim 1: Determine the efficacy of ACT for Life for preventing suicidal behavior at three- and six -months following discharge from psychiatric inpatient care. Secondary Hypotheses 1a and 1b are that ACT participants will be significantly less likely to have engaged in suicidal behavior compared to PCT participants at (a) three- and (b) six-months following discharge from psychiatric inpatient care. Secondary Aim 2: Determine the efficacy of ACT for Life for improving functioning at three-, six-, and 12-months following discharge from psychiatric inpatient care. Secondary Hypothesis 2a, 2b, and 2c are that compared to PCT participants, ACT participants will report significantly greater improvements in functioning relative to pre-treatment on the OQ-45 (a) three-, (b) six-, and (c) 12-months following discharge from psychiatric inpatient care.

Exploratory Aim: Examine candidate ACT for Life treatment mechanisms. Exploratory Hypotheses 1 and 2 are that ACT participants will show (1) greater increases from pre-treatment in psychological flexibility than PCT participants and that (2) compared to PCT participants, a greater proportion of ACT participants will engage in outpatient mental health treatment in the month following discharge from inpatient care.

The proposed RCT of ACT for Life has the potential to fill VHA's critical need for evidence-based psychotherapies that can be delivered during a typical inpatient stay, are recovery oriented, and prevent future suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for VHA care
* Currently hospitalized due to suicide risk
* Willing to be randomized and participate in either of the two conditions

Exclusion Criteria:

* Inability to provide informed consent (operationalized as inability to answer 7 questions about the study and research participants' rights)
* Inability to complete study measures or participate in treatment [based on referring clinician and study staff's judgment (e.g., due to lack of time, significant acute intoxication/withdrawal symptoms, mania, psychosis, aggression, catatonia, cognitive impairment)]
* Participation in another interventional research study
* Membership in vulnerable population (e.g., prisoner, pregnant woman)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Suicide Attempts Since Hospital Discharge Columbia-Suicide Severity Rating Scale and Medical Record Review | 3-, 6-, and 12-months post-discharge from psychiatric inpatient unit
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-administered interview that assesses for suicidal ideation and behavior based on established definitions. The C-SSRS assesses intensity of suicidal ideation, as well as actual suicide attempts, interrupted suicide attempts, and aborted suicide attempts. A combination of C-SSRS reported suicide attempts and national VHA Joint Legacy Viewer medical record review will be used to determine if participants die by suicide or engage in a suicide attempt (actual, interrupted, or aborted) during the follow-up period.
Change from Baseline on Outcome Questionnaire - 45.2 | Baseline, 1-, 3-, 6-, and 12-months post-discharge from the psychiatric inpatient unit
  The Outcome Questionnaire-45.2 (OQ-45) assesses functioning within the last week across three psychosocial domains which include symptom distress (e.g., "I feel nervous"), interpersonal relationships (e.g., "I have frequent arguments"), and social role functioning (e.g., "I find my work/school satisfying"). Sum total scores range from 0 to 180 with higher scores indicating greater symptom distress and functional impairment.

OTHER OUTCOMES:
Change from Baseline on Multidimensional Psychological Flexibility Inventory | Baseline, Pre-discharge (within 4 days of hospital discharge), and 1-, 3-, 6-, and 12-months post-discharge from psychiatric inpatient unit
  The Multidimensional Psychological Flexibility Inventory (MPFI) is a 60-item self-report measure that assesses the six dimensions of flexibility and inflexibility from ACT's psychological flexibility model, comprising ACT's theorized treatment mechanisms. Mean subscale and global composite scores range from 1 to 6 with higher scores reflecting higher levels of the dimension being assessed.
Change from Baseline on Cognitive Fusion Questionnaire - Suicidal Ideation | Baseline, pre-discharge (within 4 days of hospital discharge), and 1-, 3-, 6-, and 12-months post-discharge from psychiatric inpatient unit
  The Cognitive Fusion Questionnaire- Suicidal Ideation (CFQ-SI) is a 7-item self-report measure that assesses the extent that the respondent's behavior is impacted by suicidal thoughts. Decreases in CFQ-SI scores indicate that the respondent is better able to experience suicidal ideation without it negatively impacting their behavior. Sum scale scores can range from 7 to 49 with higher scores indicating greater fusion with suicidal ideation.
Change from Baseline on Valued Living Questionnaire | Baseline, pre-discharge (within 4 days of hospital discharge), and 1-, 3-, 6-, and 12-months post-discharge from psychiatric inpatient unit
  The Valued Living Questionnaire (VLQ) is a self-report measure that assesses participants' life values as well as their perceived success acting on those values. Participants rate the importance of ten domains of living and then rate how consistently they have lived that valued domain over the past week. The mean of the products of importance and consistency scores for each domain are calculated and can range from 1 - 100 Higher scores are desirable, indicating greater contact with values.
The Strategic Analytics for Improvement and Learning Model Post-Discharge Engagement 1 Metric | 1-month post-discharge from psychiatric inpatient unit
  The Strategic Analytics for Improvement and Learning (SAIL) Model is used to assess Veterans Health Affairs quality, safety, and value-based care. A primary SAIL metric for discharging from inpatient mental health care is the proportion of patients who engage in at least four mental health contacts within 30 days of discharge (Post-Discharge Engagement 1 Metric; PDE1). Chart review will be used to assess PDE1.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Michael Barnes, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan

IPD SHARING:
Plan to Share IPD: Yes
A final Limited Data Set will be made available, in accordance with VA policy and regulations and per compliance with current IRB and VA R&D approvals in place for this project. A study-specific DUA will be required. Data requests must be made in writing. Requests for access to data obtained from this project will be considered and responded to. Data will be provided electronically, only with a DUA in place, and per VA regulations for transferring data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After conclusion of the study and dissemination of primary and exploratory results and/or in accordance with VA policy and regulations